CLINICAL TRIAL: NCT06514573
Title: Effects of a Postbiotic Supplementation on Gastrointestinal and Core Symptoms in Autism Spectrum Disorder: A Multicenter Randomized Controlled Trial
Brief Title: Butyrate Supplementation in Children With Autism Spectrum Disorder (ASD) and Functional Gastrointestinal Disorders
Acronym: b(AUT)yrate
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Superiore di Sanità (Other)
Collaborators: University of Rome Tor Vergata (Other); Federico II University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RF-2021-12374286
Record Dates: First submitted 2024-06-26; First posted 2024-07-23 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Autism Spectrum Disorder (ASD)
Keywords: Autism Spectrum Disorder; Child; Gastrointestinal Microbiome; Microbiota; Butyrates; Fatty Acids, Volatile; Gastrointestinal Diseases; Behavioral symptoms; Gastrointestinal Symptoms; Signs and Symptoms, Digestive; Inflammatory Profile; Functional Gastrointestinal Disorders
MeSH Terms: conditions — Autism Spectrum Disorder; Gastrointestinal Diseases; Behavioral Symptoms; Signs and Symptoms, Digestive | interventions — Butyric Acid; Starch

STUDY DESIGN:
Intervention Model Description: Double-blind randomized, parallel-group, placebo-controlled study. Groups will receive oral sodium butyrate or placebo (cornstarch) for 16 weeks. The sachets and content of treatments will be indistinguishable (same color, smell, taste) and prepared by the Central Pharmacy Service of the Academic Hospital Federico II of Naples. Parents will receive an anonymous white paper box containing the sachets of placebo or butyrate, instructions for storing at room temperature, preparation (mixing the powder in water, milk, or foods), the daily amount of product, and maintaining the habitual child diet, avoiding probiotics, prebiotics, synbiotics during the entire study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinding will be maintained by making the capsules look identical. Both participants and the research staff who collect the outcome data will be blinded to treatment status. All the data will be recorded anonymously and entered into the study database by each researcher. A blinded statistician will analyze the data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Butyrate (Experimental): The butyrate groups (butyrate <=20 kg, butyrate >20 kg) will receive oral sodium butyrate (dose of 20 mg/kg body weight/daily in sachets, up to 800 mg/day maximum dose) plus ASD standard care.
  Interventions: Dietary Supplement: Sodium Butyrate
- Placebo (Placebo Comparator): The placebo groups (placebo <=20 kg, placebo >20 kg) will receive placebo (cornstarch) at the same dose and time plus ASD standard care.
  Interventions: Dietary Supplement: Placebo (cornstarch)

INTERVENTIONS:
Dietary Supplement: Sodium Butyrate — Daily supplementation with 1 sachet per day for 16 weeks
  Arms: Butyrate
Dietary Supplement: Placebo (cornstarch) — Daily supplementation with 1 sachet per day for 16 weeks
  Arms: Placebo

SUMMARY:
Autism spectrum disorder (ASD) is a neurodevelopmental condition occurring in 1:77 Italian children. Several comorbidities are reported, including functional gastrointestinal disorders (FGIDs) present in up to 70% of patients. FGIDs are disorders resulting from a combination of symptoms affecting motility, hypersensitivity, and other functions, which are not caused by anatomic or organic origin and that impact the severity of ASD core symptoms and complicate the clinical management of ASD children, especially those who are non-verbal. Evidence reports gut microbiome (GM) remodelling in ASD children, and postbiotic butyrate, a GM-derived metabolite, attenuates FGIDs in children and restores social behavior in ASD mouse models. Clinical data on butyrate effects in ASD are still scanty. The present study investigates the therapeutic effects of a 16-week oral postbiotic supplementation on clinical/behavioral profiles, gastrointestinal disturbances, gut microbiome, and immune and inflammatory biomarkers in peripheral blood and fecal samples in children with ASD and FGIDs. Using the Machine Learning (ML) approach, a subset of artificial intelligence, this study also aims to identify predictive factors implicated in the effect of the postbiotic supplementation on FGIDs, important for prevention through modulation of the microbiota. The investigators expect that treating FGIDs will have an impact on the behavioral and core symptoms of ASD and the quality of life of children and their families.

DETAILED DESCRIPTION:
ASD is a heterogeneous group of neurodevelopmental disorders with complex multifactorial etiologies requiring personalized, timely, and evidence-based interventions to improve the lives of children and their families. Medical comorbidities are common in ASD and include FGIDs, which are disorders resulting from a combination of symptoms affecting motility, hypersensitivity, and other functions, which are not caused by anatomic or organic origin. FGIDs are often associated with sleep and behavioral problems with a negative impact on clinical functioning of ASD children. Pharmacological agents that could target FGIDs in ASD children are advocated. Immune system, epigenetic, gut microbiome, mitochondrial metabolism, and gut-brain axis alterations have been implicated in ASD and FGIDs etiology and may represent potential intervention targets. The term postbiotics can be regarded as an umbrella term for all synonyms and related terms of microbial fermentation components, including many different constituents such as short-chain fatty acids, microbial cell fractions, functional proteins, extracellular polysaccharides, cell lysates, teichoic acid, peptidoglycan-derived muropeptides, and pili-type structures. Emerging data indicate that postbiotics can have direct immunomodulatory and clinically relevant effects. Evidence can be found for using postbiotics in healthy individuals to improve overall health and relieve symptoms of various diseases. In particular, the postbiotic butyrate, a Gut Microbiota-derived short-chain fatty acid, exerts protective action against FGIDs and ASD through a wide range of activities involving Gut Microbiota, immune system, epigenetic mechanisms, and mitochondrial function. Taken together, these data strongly support the hypothesis that butyrate oral supplementation can exert a therapeutic action against FGIDs and behavioral symptoms in ASD children. Butyrate has been proposed for FGIDs treatment, but its promising effect on ASD is limited to preclinical data. The present multicenter double blinded randomized controlled trial has been rigorously designed to investigate the therapeutic effects of oral butyrate supplementation in children with ASD (either idiopathic or syndromic) and FGIDs. In line with precision medicine and designing and improving diagnosis, therapeutics, and prognosis using large complex datasets, this study will implement high-performance computing and artificial intelligence in multidimensional clinical and biological datasets. The great heterogeneity of ASD, in terms of etiology and clinical presentation, requires a better understanding of who is most likely to respond to which interventions, at what intensity, and for what duration so they could be assigned to those most likely to benefit while reducing the cost of treatment to the National Health Service. Thus, there is a need to identify mediators of treatment response and moderators (factors that predict greater responsiveness to treatment, including factors that influence individuals' responses to various treatments), allowing clinicians to tailor early interventions more carefully. To this aim, mediators and moderators implicated in the effect of postbiotic supplementation on FGIDs will be explored through ML performed on clinical and biological variables collected in the digital platform Research Electronic Data Capture (REDCap). Identifying patterns/profiles of the child responding to treatment may be important in assessing risk during the early stage and planning for individualized treatment and prevention of ASD through modulation of the microbiota.

Increasing evidence suggests that the gut microbiome is one of the key modulators of gut-brain communication in ASD. The brain-gut-microbiome axis has become a compelling area of investigation in ASD, specifically in children. Previous studies suggested the presence of alteration in gut microbiome structure and function in ASD children as well as in FGIDs: decreased Bacteroidetes/Firmicutes (well-known butyrate producers) ratio in fecal samples of ASD children and significantly reduced butyrate level production by the gut microbiome of ASD children.

Butyrate is a widely known histone deacetylase inhibitor due to its ability to cross the blood brain barrier. Previous research has shown that treatment with oral sodium butyrate improved behavioral deficits in BTBR mice, one of the most robust animal models of ASD. The gene expression analyses of the frontal cortex revealed that the effects of butyrate on behavior were attributable to a positive modulation of genes involved in excitatory/inhibitory balance and neuronal activation. Specifically, sodium butyrate downregulated the neuronal activation marker genes and upregulated the inhibitory neurotransmitter genes. In addition, a double-blind trial in 3-8 year old children with ASD was recently conducted to assess the effect of L. Reuteri supplementation (6 months) on social deficits, gastrointestinal (GI) symptoms, and immune response. Unpublished findings showed that L. Reuteri significantly increased scores of Adaptive Behavior Assessment System social subdomains and decreased the total score of the Social Responsiveness Scale and gastrointestinal (GI) symptoms at 6 months. Behavioral results based on intelligent quotient (IQ) stratification also revealed the L. Reuteri efficacy on social and GI domains in ASD children with normal IQ range. These studies highlight the promising role of probiotics and postbiotics in ASD children.

Aims. A multicenter, double-blind, sequential Randomized Controlled Trial of butyrate vs placebo will be carried out in 128 ASD children (estimated sample size) to evaluate the efficacy of the postbiotic supplementation on functional gastrointestinal disorders in children with ASD. A secondary aim is to define whether and to what extent the butyrate supplementation could influence ASD behavioral and core symptoms. The third aim is to identify clinical and/or biological determinants of ASD children's response to postbiotic supplementation.

Materials and Methods. Azienda Ospedaliera Universitaria Federico II of Naples and Policlinico Tor Vergata Hospital will invite parents of 3-6 years old ASD children to participate in the study. If they agree, full information about the protocol will be provided and written signed informed consent will be collected. ASD diagnosis, severity, and clinical functioning will be defined according to Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria and gold-standard tests; the FGIDs diagnosis will be performed using the Rome III Criteria questionnaire, and the 6-GSI. Children's dietary habits will be assessed by the 3-day food diary. Clinical centers will send age, gender, and IQ data to Istituto Superiore di Sanità for the centralized randomization procedure in the REDCap platform. At baseline (Timepoint 0), parents will be invited to Azienda Ospedaliera Universitaria Federico II of Naples and Policlinico Tor Vergata Hospital for a comprehensive clinical evaluation including anamnestic interview and the administration of standardized tests for autism and gastrointestinal symptoms, global development and adaptive and behavioral functioning. Blood and faecal samples for genetic and metabolic analysis will be collected, and electroencephalography will also be performed.

Parents will receive butyrate or placebo supplementation for 16 weeks (4 months), according to the allocation process. Treatment will be numbered according to the randomization scheme with no reference to group assignment, only known by the Istituto Superiore di Sanità statistician who generates the list. The Central Pharmacy Service of the Academic Hospital Federico II of Naples will prepare the sachets and indistinguishable (same color, smell, taste) treatments' content. Clinical centers will repeat a full evaluation at the end of the supplementation period (Timepoint 1). At Timepoint 2 (after 4 months by the end of Timepoint 1), parents will be asked to fill Timepoint 1 questionnaires to evaluate the long-term effect - consolidation - of supplementation. To avoid further discomfort to children and families, blood and fecal sampling will not be collected at Timepoint 2.

Determinants of response to the butyrate supplementation and biomarkers that differentiate responders from non-responders will be identified by implementing high-performance computing and artificial intelligence to the multidimensional clinical and biological datasets collected in the digital platform developed and managed by Istituto Superiore di Sanità. Using the ML approach, a subset of artificial intelligence, the University Federico II of Naples will analyze the dataset to establish relationships without preassigned modeling. ML is an innovative approach to provide robust predictions, overcoming descriptive statistical models, and proving a digital twin for the considered phenomena. Clinical, behavioral, inflammatory, and immunological factors are altered in ASD. However, the great variability among individuals with ASD of these problems makes it difficult to predict who is most likely to respond to a specific intervention, at what intensity, and for what duration. To this aim, the investigators will develop a probabilistic multi-domain data integration model consisting of the gut microbiome, immune, and inflammatory biomarkers in peripheral blood and fecal samples, and clinical/behavioral biomarkers using ML to improve therapeutics and predict the prognosis of ASD. Clinical and behavioral variables to be included in the dataset will be collected through the tests/questionnaires described in the experimental design. Gut microbiome, immune and inflammatory variables will be gathered on blood and fecal samples at baseline (Timepoint 0) and at the end of supplementation (Timepoint 1). The composition of the gut microbiome will be characterized by shotgun metagenomics. Genomes of dominant strains will also be reconstructed with a recently validated standard pipeline and compared to define if a strain-level variation exists upon treatment with butyrate. Fecal Short-Chain Fatty Acids (SCFAs: acetate, propionate, and butyrate) levels will be determined by gas chromatograph-mass spectrometry, as previously described. Altered composition of the gut microbiome may alter the gut barrier, potentially allowing the translocation of bacteria and their antigens, toxins, and metabolites and result in multiple alterations of cytokines' production, immune cell populations, as well as cellular activation markers.

Randomization and allocation concealment will be performed by the Istituto Superiore di Sanità. Randomization will be generated using the procedure Ralloc in STATA, managed through the RECap platform after enrollment and provided to clinicians by the Istituto Superiore di Sanità. Specific standard operative procedures (SOPs) were defined to garantee study and trial integrity. A blinded statistician will analyze data using Stata 16.1.

ELIGIBILITY:
Inclusion Criteria:

* children aged 3-6 years
* both sexes
* ASD diagnosis and presence of FGIDs (6-item Gastrointestinal Severity Index (6-GSI) >7 from > 3 months)

Exclusion Criteria:

* age 6 years
* uncertain FGIDs diagnoses
* FGIDs symptoms duration <3 months
* concomitant presence of other chronic condition (adverse food reactions, metabolic disorders, infections)
* malformation and Gi or urinary tracts chronic diseases
* immunodeficiencies
* diabetes
* neurologic/cardiovascular/autoimmune diseases
* obesity
* malnutrition
* antibiotics and/or pre-/pro-/synbiotics use 6 months prior to enrollment
* last 12 months participation into other clinical trials

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 128 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Gastrointestinal symptom severity. | At baseline (Timepoint 0) and at 4 months (Timepoint 1)
  Rate of subjects presenting a clinically relevant improvement in Functional Gastrointestinal Disorders (FGIDs) severity, measured by 6-item Gastrointestinal Severity Index (6-GSI) score decrease >4 points.
  The Gastrointestinal Severity Index (6-GSI) score is the sum of the individual item scores.
  The higher it is, the worse is the outcome. Score range for each item: 0, 1, 2 (0 no symptoms, 1 mild symptoms, 2 severe symptoms).

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | At 4 months (Timepoint 1) and at 8 months (Timepoint 2)
  Parental questionnaires on the presence of nausea, skin irritation, itching, patches on the skin, stomach ache, flatulence, meteorism, vomiting, constipation, increased/decreased appetite, heartburn, reflux, burping.
  Measured in hours or days of symptoms' duration.
Unexplained daytime irritability | At 4 months (Timepoint 1) and at 8 months (Timepoint 2)
  Parental questionnaires on the presence of angry outbursts, bouts of crying, easy frustration, mood swings, aggression, restlessness.
  Measured by symptom intensity during daytime: light, mild, severe.
Nocturnal awakening | At 4 months (Timepoint 1) and at 8 months (Timepoint 2)
  Parental questionnaires on the presence of night waking. Measured as Yes (number of episodes) or No.
Persistency of Functional Gastrointestinal Disorders severity improvement | At 4 months (Timepoint 1) and at 8 months (Timepoint 2)
  Measured by 6-item Gastrointestinal Severity Index (6-GSI) score: the sum of the individual item scores.
  The higher it is, the worse is the outcome. Score range for each item: 0, 1, 2 (0 no symptoms, 1 mild symptoms, 2 severe symptoms).
Gut Microbiota structure and function (fecal Short-Chain Fatty Acids levels, SCFAs) | At baseline (Timepoint 0) and at 4 months (Timepoint 1)
  Bacterial DNA extraction from one fecal sample will be carried out by shotgun metagenomics. Fecal SCFAs (acetate, propionate and butyrate) levels will be measured using the second fecal sample by gas chromatograph-mass spectrometry and expressed in mM (millimolar) with a range of 0-∞.
Changes in Autism Spectrum Disorder severity | At baseline (Timepoint 0), at 4 months (Timepoint 1) and 8 months (Timepoint 2)
  Measured by Social Responsiveness Scale-2 (SRS-2). Score range for each item: 0-100. The higher the score, the worse the outcome.
Changes in Autism Spectrum Disorder behavior | At baseline (Timepoint 0), at 4 months (Timepoint 1) and 8 months (Timepoint 2)
  Measured by Aberrant Behavior Checklist (ABC). Score range for each item: 0-999. The higher the score, the worse the outcome.
Changes in Autism Spectrum Disorder symptomatology: repetitive behaviors | At baseline (Timepoint 0), at 4 months (Timepoint 1) and 8 months (Timepoint 2)
  Delta of scores at Repetitive Behavior Scale-Revised (RBS-R), a 43-item scale. Score range for each item: 0-100. Higher scores are related to greater severity of symptoms.
Changes in Sensory input reaction | At baseline (Timepoint 0), at 4 months (Timepoint 1) and 8 months (Timepoint 2)
  Measured by Sensory Profile 2 (SP-2) scores. Score range for raw score: 86-430. Score range for percentiles: 0-100. The further away from the mean score, the more pathological.
  Score categories for sensitivity level: 1,2,3,4,5.
  1. Severe hyposensitivity (< -2 Standard Deviation)
  2. Mild hyposensitivity (between -1 e -2 Standard Deviation)
  3. Typical sensitivity (between -1 and 1 Standard Deviation)
  4. Mild hypersensitivity (between 1 and 2 Standard Deviation)
  5. Severe hypersensitivity (> 2 Standard Deviation)
Changes in Adaptive Functioning | At baseline (Timepoint 0), at 4 months (Timepoint 1) and 8 months (Timepoint 2)
  Measured by Vineland Adaptive Behavior Scales-II (VABS-II). Score range for each item: 0-160. The higher the score, the better the outcome.
Changes in emotional/behavioral problems | At baseline (Timepoint 0), at 4 months (Timepoint 1) and 8 months (Timepoint 2)
  Measured by Child Behavior Checklist (CBCL syndrome subscales). Score range for each item: 0-999. The higher the score, the worse the outcome.
Changes in sleep disorders | At baseline (Timepoint 0), at 4 months (Timepoint 1) and 8 months (Timepoint 2)
  Measured by Children's Sleep Habits Questionnaire Abbreviated (CSHQ).
  Score ranges for items:
  Bedtime (0-63), Sleep behavior (0-49), Waking during the night (0-14), Morning wake up (0-28).
  Total sleep disturbance score: the sum of the individual item scores (0-154). The higher the score, the worse the outcome.
Sleep disturbance assessment | At baseline (Timepoint 0), at 4 months (Timepoint 1) and 8 months (Timepoint 2)
  Measured by Sleep Disturbance Scale for Children (SDSC).
  Score ranges for items:
  Sleep onset and maintenance disorders (7-35), Sleep breathing disorders (3-15), Arousal disorders (3-15), Wake-Sleep Transition Disorder (6-30), Excessive sleepiness disorder (5-25), Nocturnal hyperhidrosis (2-10).
  Total score: the sum of the individual item scores (26-130). Higher scores indicate more acute sleep disturbances.
Impact on parental quality of life | At baseline (Timepoint 0), at 4 months (Timepoint 1) and 8 months (Timepoint 2)
  Evaluated through the Quality of life questionnaire (EUROHIS QOL-8). Score range for each item: 1-5. Higher score indicates a better condition. Overall index score: the mean of the individual scores, ranging from 1 to 5 with a higher score indicating a better quality of life.
Serum proinflammatory and regulatory cytokines | At baseline (Timepoint 0) and at 4 months (Timepoint 1)
  Intracellular expression of cytokines (IL-1beta, IL-5, IL-6, IL-10, IL-15, IL-17, TGF-beta, TNF-alpha, IFN-alpha, IFN-gamma) measured by Enzyme-Linked Immuno Assay (ELISA).
  All reported as pg/ml.
Plasmatic levels of chemochines involved in the migration of inflammatory cells within the CNS (Part 1) | At baseline (Timepoint 0) and at 4 months (Timepoint 1)
  Expression of ICAM-1, PECAM-1, and P-selectin measured by Enzyme-Linked Immuno Assay (ELISA).
  All reported as ng/ml.
Plasmatic levels of chemochines involved in the migration of inflammatory cells within the CNS (Part 2) | At baseline (Timepoint 0) and at 4 months (Timepoint 1)
  Expression of L-selectin measured by Enzyme-Linked Immuno Assay (ELISA). Reported as pg/ml.
Peripheral blood mononuclear cells features (Part 1) | At baseline (Timepoint 0) and at 4 months (Timepoint 1)
  Characterization of peripheral blood mononuclear cells immunophenotype by flow cytometry (Cytoflex, Beckman Coulter).
  All expressed in % (range 0,000-100,000):
  Lymphocytes, Monocytes, Granulocytes,CD3, CD4, CD8, CD19, CD16, CD56, HLA-DR Monocytes, HLA-DR Lymphocytes, HLADRMONOLYMPH, CD169Leukocytes, CD169Lymphocytes, CD169Monocytes, CD169Granulocytes, HLADRLLeukocytes, HLADRLymphocytes, HLADRMonocytes, HLADRGranulocytes, HLADRCD169Leukocytes, HLADRCD169Lymphocytes, HLADRCD169Monocytes, HLADRCD169Granulocytes, CD3_tube2, CD4_tube2, CD4CM, CD4NAIVE, CD4EM, CD4TEM, CD8_tube2, CD8CM, CD8NAIVE, CD8EM, CD8TEM, CD4PD1CD57, CD4CD57, CD4PD1, CD8PD1CD57, CD8CD57, CD8PD1, CD19_tube2, Marginal, NaiveB, IgDmCD27m, IgDmCD27p, CD21lowCD38low, IgMpIgDp, IgMmIgDp, IgDmIgMm, IgMpIgDm, IgMpCd27pCD38p, Unswitchedmemory, IgMpCD27mCD38dim, IgMpCD27mCD38high, IgDmIgMmCD27pCD38high, Switchedmemory, IgMmIgDmCD27mCD38low, IgMmIgDmCD27mCD38high, Plasmablasts, IgMpCD27m, TransitionalBcells
Peripheral blood mononuclear cells features (Part 2) | At baseline (Timepoint 0) and at 4 months (Timepoint 1)
  Characterization of peripheral blood mononuclear cells immunophenotype by flow cytometry (Cytoflex, Beckman Coulter).
  All expressed as absolute number/ml:
  CD169MEDLYMPH, CD169MEDMONO, CD64MEDLYMPH, CD64MEDNEUTRO
Peripheral blood mononuclear cells features (Part 3) | At baseline (Timepoint 0) and at 4 months (Timepoint 1)
  Characterization of peripheral blood mononuclear cells immunophenotype by flow cytometry (Cytoflex, Beckman Coulter).
  All expressed as Ratio, absolute number:
  CD169 Monocytes/Lymphocytes RMFI, CD64 Neutrophils/Lymphocytes RMFI

CONTACTS AND LOCATIONS:
Overall Officials: Maria Luisa Scattoni, Ph.D., Principal Investigator — Istituto Superiore di Sanità
Locations (3):
- Italy (3):
  - Azienda Ospedaliera Universitaria Federico II, Naples
  - Policlinico Tor Vergata Hospital, Rome
  - Istituto Superiore di Sanità, Rome

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saurman V, Margolis KG, Luna RA. Autism Spectrum Disorder as a Brain-Gut-Microbiome Axis Disorder. Dig Dis Sci. 2020 Mar;65(3):818-828. doi: 10.1007/s10620-020-06133-5. PMID 32056091
- [Background] Zheng Y, Verhoeff TA, Perez Pardo P, Garssen J, Kraneveld AD. The Gut-Brain Axis in Autism Spectrum Disorder: A Focus on the Metalloproteases ADAM10 and ADAM17. Int J Mol Sci. 2020 Dec 24;22(1):118. doi: 10.3390/ijms22010118. PMID 33374371
- [Background] Coretti L, Paparo L, Riccio MP, Amato F, Cuomo M, Natale A, Borrelli L, Corrado G, Comegna M, Buommino E, Castaldo G, Bravaccio C, Chiariotti L, Berni Canani R, Lembo F. Gut Microbiota Features in Young Children With Autism Spectrum Disorders. Front Microbiol. 2018 Dec 19;9:3146. doi: 10.3389/fmicb.2018.03146. eCollection 2018. PMID 30619212
- [Background] Liu J, Gao Z, Liu C, Liu T, Gao J, Cai Y, Fan X. Alteration of Gut Microbiota: New Strategy for Treating Autism Spectrum Disorder. Front Cell Dev Biol. 2022 Mar 3;10:792490. doi: 10.3389/fcell.2022.792490. eCollection 2022. PMID 35309933
- [Background] Wei L, Singh R, Ro S, Ghoshal UC. Gut microbiota dysbiosis in functional gastrointestinal disorders: Underpinning the symptoms and pathophysiology. JGH Open. 2021 Mar 23;5(9):976-987. doi: 10.1002/jgh3.12528. eCollection 2021 Sep. PMID 34584964
- [Background] Canani RB, Costanzo MD, Leone L, Pedata M, Meli R, Calignano A. Potential beneficial effects of butyrate in intestinal and extraintestinal diseases. World J Gastroenterol. 2011 Mar 28;17(12):1519-28. doi: 10.3748/wjg.v17.i12.1519. PMID 21472114
- [Background] Rose S, Bennuri SC, Davis JE, Wynne R, Slattery JC, Tippett M, Delhey L, Melnyk S, Kahler SG, MacFabe DF, Frye RE. Butyrate enhances mitochondrial function during oxidative stress in cell lines from boys with autism. Transl Psychiatry. 2018 Feb 2;8(1):42. doi: 10.1038/s41398-017-0089-z. PMID 29391397
- [Background] Scattoni ML, Gandhy SU, Ricceri L, Crawley JN. Unusual repertoire of vocalizations in the BTBR T+tf/J mouse model of autism. PLoS One. 2008 Aug 27;3(8):e3067. doi: 10.1371/journal.pone.0003067. PMID 18728777
- [Background] Turriziani L, Ricciardello A, Cucinotta F, Bellomo F, Turturo G, Boncoddo M, Mirabelli S, Scattoni ML, Rossi M, Persico AM. Gut mobilization improves behavioral symptoms and modulates urinary p-cresol in chronically constipated autistic children: A prospective study. Autism Res. 2022 Jan;15(1):56-69. doi: 10.1002/aur.2639. Epub 2021 Nov 23. PMID 34813183
- [Background] Adams JB, Johansen LJ, Powell LD, Quig D, Rubin RA. Gastrointestinal flora and gastrointestinal status in children with autism--comparisons to typical children and correlation with autism severity. BMC Gastroenterol. 2011 Mar 16;11:22. doi: 10.1186/1471-230X-11-22. PMID 21410934
- [Background] Pasolli E, Truong DT, Malik F, Waldron L, Segata N. Machine Learning Meta-analysis of Large Metagenomic Datasets: Tools and Biological Insights. PLoS Comput Biol. 2016 Jul 11;12(7):e1004977. doi: 10.1371/journal.pcbi.1004977. eCollection 2016 Jul. PMID 27400279
- [Background] De Filippis F, Paparo L, Nocerino R, Della Gatta G, Carucci L, Russo R, Pasolli E, Ercolini D, Berni Canani R. Specific gut microbiome signatures and the associated pro-inflamatory functions are linked to pediatric allergy and acquisition of immune tolerance. Nat Commun. 2021 Oct 13;12(1):5958. doi: 10.1038/s41467-021-26266-z. PMID 34645820
- [Background] Lopez-Cacho JM, Gallardo S, Posada M, Aguerri M, Calzada D, Mayayo T, Lahoz C, Cardaba B. Characterization of immune cell phenotypes in adults with autism spectrum disorders. J Investig Med. 2016 Oct;64(7):1179-85. doi: 10.1136/jim-2016-000070. Epub 2016 Jun 13. PMID 27296457
- [Background] Horiuchi F, Yoshino Y, Kumon H, Hosokawa R, Nakachi K, Kawabe K, Iga JI, Ueno SI. Identification of aberrant innate and adaptive immunity based on changes in global gene expression in the blood of adults with autism spectrum disorder. J Neuroinflammation. 2021 Apr 30;18(1):102. doi: 10.1186/s12974-021-02154-7. PMID 33931079
- [Background] Kim E, Paik D, Ramirez RN, Biggs DG, Park Y, Kwon HK, Choi GB, Huh JR. Maternal gut bacteria drive intestinal inflammation in offspring with neurodevelopmental disorders by altering the chromatin landscape of CD4+ T cells. Immunity. 2022 Jan 11;55(1):145-158.e7. doi: 10.1016/j.immuni.2021.11.005. Epub 2021 Dec 7. PMID 34879222
- [Background] Bourgoin P, Biechele G, Ait Belkacem I, Morange PE, Malergue F. Role of the interferons in CD64 and CD169 expressions in whole blood: Relevance in the balance between viral- or bacterial-oriented immune responses. Immun Inflamm Dis. 2020 Mar;8(1):106-123. doi: 10.1002/iid3.289. Epub 2020 Feb 7. PMID 32031762
- [Background] Minutolo A, Petrone V, Fanelli M, Iannetta M, Giudice M, Ait Belkacem I, Zordan M, Vitale P, Rasi G, Sinibaldi-Vallebona P, Sarmati L, Andreoni M, Malergue F, Balestrieri E, Grelli S, Matteucci C. High CD169 Monocyte/Lymphocyte Ratio Reflects Immunophenotype Disruption and Oxygen Need in COVID-19 Patients. Pathogens. 2021 Dec 18;10(12):1639. doi: 10.3390/pathogens10121639. PMID 34959594
- [Background] Drossman DA. Rome III: the new criteria. Chin J Dig Dis. 2006;7(4):181-5. doi: 10.1111/j.1443-9573.2006.00265.x. PMID 17054578